CLINICAL TRIAL: NCT00689910
Title: Pharmacokinetics of Raltegravir During Third Trimester Pregnancy and Post-Partum
Status: Withdrawn | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Francesca Aweeka, University of California, San Francisco
Other Study IDs: PK of Ral in Pregnant Women
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infections
Keywords: pharmacokinetics; pregnancy; Raltegravir; HIV; antiretroviral; Treatment of HIV in pregnant women with Raltegravir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Cervicovaginal lavage fluid Endocervical canal fluid

SUMMARY:
This study will evaluate the pharmacokinetic disposition of raltegravir in pregnant HIV-1 infected women. These results will be compared to pharmacokinetic data obtained following pregnancy as well as to studies previously carried out in nonpregnant women and male patients. By determining the disposition characteristics for this specific patient population, antiretroviral (ARV) dosing can be optimized during pregnancy. Appropriate dosing is necessary to minimize adverse effects, slow progression of disease, and further reduce the risk for vertical transmission. Data will also be obtained on genital tract penetration and placenta transfer of raltegravir to the newborn.

The subjects enrolled in this study will take an antiretroviral based regimen containing raltegravir twice daily both during and after their pregnancy. The specific regimen will be chosen by their own primary care provider based on their antiretroviral history and resistance testing. They will undergo a series of blood sampling for pharmacokinetic analysis over 12 hours on two occasions; a) during their 3rd trimester and b) approximately 3 months postpartum. Concentrations of raltegravir in the infant will be assessed by cord and infant blood sample at delivery and a blood sample at approximately 3 months of age.

Hypothesis: The pharmacokinetic exposure of raltegravir as measured by the 12 hour area under the plasma concentration versus time curve (AUC0-12h) during third trimester pregnancy is similar to the AUC0-12h estimated three months post-partum.

ELIGIBILITY:
Inclusion Criteria:

* Female, 16 years old or older
* Pregnant, at least 14 weeks gestation in order to initiate raltegravir treatment if decided by their pregnancy health care provider. The first pharmacokinetic study visit occurs no sooner than 26 weeks gestation (3rd trimester)
* Normal fetal heart motion by ultrasound, vital signs and brief physical exam as conducted by their primary pregnancy health care provider within two weeks of study entry (part of their standard prenatal care)
* Intolerance or resistance to at least two classes of antiretroviral agents
* Availability of a raltegravir-optimized background regimen based on referring provider's selection and resistance testing
* English or Spanish speaking

Exclusion Criteria:

* Inability to follow study protocol or drug administration
* Women who are planning to breastfeed (this is not recommended for HIV-infected women to reduce HIV transmission to the baby)
* Women unable to sign informed consent
* Women with a history of anaphylaxis or other life threatening adverse event associated with antiretroviral therapy

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preliminary eligibility will be determined by the study investigators, research staff, and the patient's primary pregnancy healthcare provider. During a dedicated visit to the primary investigator's office, potential participants will undergo a screening examination including review of physical exam and blood work obtained by their primary pregnancy provider within two weeks of study enrollment. Those that qualify will then provide written consent and be able to continue in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - East Bay AIDS Center, Oakland, California
  - UC Davis, Sacramento, California
  - San Francisco General Hospital, San Francisco, California
  - UC San Francisco, San Francisco, California